CLINICAL TRIAL: NCT00936416
Title: Assessment of Renal Physiology (Glomerular Filtration Rate and Blood Flow) by MRI With Validation by Inulin and Para-Aminohippuric Acid Clearance in Normal Volunteers
Brief Title: Assessment of Renal Physiology by Magnetic Resonance Imaging (MRI) in Normal Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Kartik Jhaveri, MD/Principal Investigator, University Health Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UHN09-0096B
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Glomerular Filtration Rate; Renal Blood Flow
Keywords: Glomerular Filtration Rate; Renal Blood Flow; MRI; Inulin; Para-Aminohippuric Acid
MeSH Terms: interventions — Inulin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GFR and RBF followed by MRI (Experimental): Subjects will undergo GFR and renal blood flow estimation by Inulin and PAH clearance method, followed by a MRI test. The MRI examination will be performed on the same day as the inulin/PAH procedure.
  Interventions: Procedure: Inulin and PAH clearance and MRI

INTERVENTIONS:
Procedure: Inulin and PAH clearance and MRI — GFR and renal blood flow estimation by Inulin and PAH clearance will be performed in the Renal Physiology Lab for approximately 2.5 hours;
  The MRI test will be performed afterwards at Medical Imaging department and last about 45 minutes.

SUMMARY:
Estimation of Glomerular Filtration Rate (GFR) is the primary test used to assess patients with renal disease. Although serum creatinine based GFR and nuclear medicine based estimations are routinely used in clinical practice, GFR estimation by Inulin is the recommended gold standard. Inulin based estimation of GFR is cumbersome and time consuming.

A decrease in blood flow to the kidney (Renal Blood Flow (RBF)) is known to cause a decrease in GFR. RBF is typically determined using radioactive tracers, contrast MRI or a cumbersome para-aminohippuric acid (PAH) clearance method.

MRI based assessment of GFR and RBF have been suggested to provide reasonable accuracy. Most of these studies did not compare the GFR and RBF estimation directly to Inulin and PAH clearance which are ther gold standards . In this study we propose to estimate MRI based GFR estimation directly to Inulin and noncontrast MRI based derived RBF to PAH to assess if MRI is an accurate test of kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers with no known renal disease
* Ages between 18-65 years
* Normal routine urinalysis
* Estimated GFR (eGFR) >=90mls/min
* Arterial pressure < 130/85
* No medications (birth control pills and vitamins are acceptable)

Exclusion Criteria:

* Pregnancy
* Age <18y or >65y
* Proteinuria or hematuria as determined by routine urinalysis
* Estimate GFR (eGFR) < 90 ml/min
* Known history or requirement of treatment for hypertension
* Known allergy to inulin or PAH
* MRI contrast allergy, general contraindications to MRI such as pacemaker, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
GFR estimation comparison between results obtained by MRI and Inulin clearance method. Blood flow estimation comparison between results obtained by MRI and PAH clearance method. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Jhaveri, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada